CLINICAL TRIAL: NCT02989831
Title: The Effects of Random Vibrations on the Vibratory Perception Threshold of the Foot and Standing Balance in People With Diabetic Neuropathy
Brief Title: The Effect of Random Vibrations on Perception and Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Juha M Hijmans, PhD, University Medical Center Groningen
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: NL48517.042.14
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Neuropathy
Keywords: diabetic neuropathy; foot ulcers; random vibration; vibration perception threshold; mechanical noise
MeSH Terms: conditions — Diabetic Neuropathies; Foot Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vibrating insoles 'on' (Experimental): Duration: 30-60 seconds
  Interventions: Device: Vibrating insoles 'on'
- Vibrating insoles 'off' (No Intervention): Duration: 30-60 seconds

INTERVENTIONS:
Device: Vibrating insoles 'on' — Duration: 30-60 seconds
  Arms: Vibrating insoles 'on'

SUMMARY:
The purpose of this study is to investigate the effects of vibrating insoles on vibration perception threshold (VPT) and balance of people with diabetic neuropathy.

DETAILED DESCRIPTION:
Rationale: People with diabetes mellitus often suffer from polyneuropathy. Reduced somatosensation of the feet due to polyneuropathy is one of the major risk factors for ulceration at the plantar side of the feet and may often cause problems in balance. It has been shown that the application of a mechanical noise signal to the feet (a vibration with a random frequency) can reduce the sensation threshold and improve standing balance. However, techniques used in research so far have several problems that limit applicability in daily practice. New vibrating insoles have been developed that overcome these problems, but it is unknown if these insoles have the same effects.

Study population: Two samples of 20 consecutive patients with diabetes mellitus will be included. Patients will be included if their VPT is between 25 and 45V. Patients with a history of ulceration on MTP, halllux or heel region will be included in the first sample group. In the second sample group patients with no history of ulceration will be included. Patients with an ulceration or (a history of) amputation will be excluded in both groups.

Intervention: First, participants will be standing on vibrating insoles placed on a platform for the measurement of VPT. Secondly, participants will be standing on a force platform while wearing standardized shoes in which vibrating insoles are placed. The insoles are either turned on (i.e. random vibrations applied) or off (i.e. no random vibrations applied).

Main study parameters: Vibration perception threshold and centre of pressure displacements.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus, type I or type II
* Aged 18 years or older
* Diagnosed with neuropathy
* VPT between 25-45V
* Understand Dutch or English
* Is able to detect the stimulus at full power

Exclusion Criteria:

* A history of neuropathic conditions other than diabetes mellitus
* Problems with the somatosensory or motor system that affect balance or plantar sensation, not related to DM (for example: CVA)
* Severe visual problems
* Current ulcer
* (a history of) amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Decrease in Vibration Perception Threshold (VPT) due to vibrating insoles | One minute
Difference in center of pressure displacement (balance) between the two conditions. | 1 minute

SECONDARY OUTCOMES:
Difference in mediolateral velocity of the centre of pressure displacement between the two conditions (vibrating insoles 'on' or 'off'). | 1 minute
Difference in anteroposterior velocity of the centre of pressure displacements between the two conditions (insoles 'on' or 'off') | 1 minute

CONTACTS AND LOCATIONS:
Overall Officials: Juha M Hijmans, PhD, Principal Investigator — Center for Rehabilitation, UMCG

IPD SHARING:
Plan to Share IPD: No